CLINICAL TRIAL: NCT01423708
Title: Terapia Con Everolimus Nel Trapianto de Novo di Fegato: Uno Studio Multicentrico Randomizzato
Brief Title: Everolimus in de Novo Liver Transplantation: a Multicentre Randomized Study
Acronym: EPOCAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Director of the Hepatobiliary Surgery and Liver Transplantation Unit, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1956P; 2009-016176-78 (EudraCT Number)
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Liver Failure; Liver Diseases; Liver Cirrhosis; Liver Neoplasms
Keywords: Liver Transplantation; Graft Rejection; Graft Survival; Transplantation Immunology; Anti-Rejection Therapy; Immunosuppression; Organ Transplantation; Host vs Graft Reaction; Gastroenterology; Hepatology
MeSH Terms: conditions — Liver Failure; Liver Diseases; Liver Cirrhosis; Liver Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard immunosuppression protocol with Tacrolimus, maintaining trough levels between 6 and 12 ng/ml in the first month, in association with steroids (20 mg/day with subsequent weaning within 3 months after transplantation).
- Everolimus (Experimental): Administration of Everolimus in association with Tacrolimus and steroids.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Administration of Everolimus within 24 hours from the time of randomization (7 days from the time of transplantation) in association with Tacrolimus and steroids. The first dose level of the trough will be performed at day 7 after initiation of therapy. After the reaching an Everolimus trough level of >5ng/ml (final target 6-12 ng/ml), there will be a gradual weaning of tacrolimus (bringing Tacrolimus blood levels <5 ng/ml) with discontinuation of Tacrolimus within 30 days after transplantation when possible.
  Other Names: Certican; Afinitor; Zortress
  Arms: Everolimus

SUMMARY:
Safety and Efficacy of Everolimus in adult de novo liver transplant recipients.

DETAILED DESCRIPTION:
This prospective study was designed to evaluate the feasibility and effectiveness of the use of Everolimus in the minimization and possible suspension of calcineurin inhibitors in adult liver transplant patients. The study will take into account a control group (standard immunosuppression with tacrolimus and steroids) after induction with anti-IL2 Antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 70 years of age,
* Patients undergoing de novo liver transplantation from cadaveric donor with a functional graft at the time of randomization,
* Transplantation from cadaveric donor whole or split liver,
* Patients able to communicate properly with the study investigators, to understand and respond to the needs of the protocol and who have given written consent
* Cold ischemia time <12 hours

Exclusion Criteria:

* Physical or laboratory abnormalities or mental illness within 2 weeks before randomization such that, in the opinion of the investigator, may interfere with participation in the study
* Women who are pregnant (positive test with hCG values> 5mUI/ml) or breast-feeding
* Women of childbearing potential, with the following exceptions: a) women in menopause (spontaneous amenorrhea for at least 12 months, spontaneous amenorrhea for at least 6 months with FSH levels >40 mIU/ml, surgical bilateral oophorectomy at least 6 weeks before baseline, with or without hysterectomy) b) women who use one or more reliable and approved methods of contraception for the duration of the study and for the three months following discontinuation of study treatment.
* Patients who undergo transplantation or multivisceral transplantation of pancreatic islets, or who have previously undergone organ transplantation or tissue.
* Patients who undergo combined liver-kidney transplantation
* Patients who undergo living donor liver transplantation
* Patients who undergo ABO-incompatible liver transplantation
* Patients who undergo transplantation from donors positive for HBV surface antigen or HIV
* History of malignant disease at any site in the 3 year period prior, regardless of whether or not there is evidence of recurrence or metastasis. (Except non-metastatic skin cancers such as basal cell or squamous cell carcinoma of the skin, or hepatocellular carcinoma)
* Patients receiving other investigational drugs within 4 weeks before baseline or who are currently enrolled in other clinical trials
* Patients who show hypersensitivity to the drug (or drugs similar to Everolimus - Former macrolides) or class or pharmaceutical excipients. Also, when there are contraindications
* A history of coagulopathy or the presence of any medical condition that requires long-term anticoagulant therapy after transplantation (The use of low-dose ASA is admissible)
* Platelet count <=40.000/mm3 or WBC count <2000/mm3 or hemoglobin <=7g/dl at the time of randomization
* Severe systemic infections
* High cholesterol levels (>350mg/dl) or severe hypertriglyceridemia (>500mg/dl). Patients with compensated hyperlipidemia are eligible.
* Diagnosis of pre-transplant autoimmune liver disease (PBC, sclerosing cholangitis)
* Acute Liver Failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2010-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Biopsy-proven rejection episodes (BPAR) | 3 months
Graft survival | 3 months
Patient post-Liver Transplantation survival | 3 months
Everolimus monotherapy | 30 days
  Patients not requiring calcineurin inhibitors (CNI)

SECONDARY OUTCOMES:
Renal function evaluation | 24 months
  Impact of therapy on renal function, evaluated by creatinine clearance according to the Modification of Diet in Renal Disease (MDRD) Study.
Requests for dialysis | 24 months
Incidence of Adverse Events | 24 months
  Evaluation of common post Liver Transplantation Adverse Events:
  wound healing, bone marrow depression, hyperlipidemia, proteinuria, diabetes mellitus, diagnosed hypertension, infections, levels of HCV.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, MD, Study Chair — Azienda Ospedaliera di Padova
Locations (7):
- Italy (7):
  - Ospedali Riuniti - Bergamo, Bergamo, BG
  - Irccs Ospedale Maggiore Policlinico Di Milano, Milan, MI
  - Ospedale Ca' Granda-Niguarda - Milano, Milan, MI
  - Azienda Ospedaliera di Padova, Padua, PD
  - Policlinico Universitario Gemelli Di Roma, Roma, RM
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino, Torino, TO
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, UD

REFERENCES:
- See also: Hepatobiliary surgery and Liver Transplantation Unit, University Hospital of Padua (Italy) — http://www.fegatochirurgia.com/